CLINICAL TRIAL: NCT02512640
Title: Comparison of Oxidative Stress Changes in Different Ventilation Strategies During Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CGMH-IRB-102-0112A3
Record Dates: First submitted 2015-07-06; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Reperfusion Injury; Oxidative Stress
Keywords: Pressure-controlled ventilation; Volume-controlled ventilation; Laparoscopy; Oxidative stress
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volume-controlled ventilation (Active Comparator): Volume-controlled ventilation throughout the surgery
  Interventions: Procedure: Volume-controlled ventilation
- Pressure-controlled ventilation (Active Comparator): Pressure-controlled ventilation throughout the surgery
  Interventions: Procedure: Pressure-controlled ventilation

INTERVENTIONS:
Procedure: Volume-controlled ventilation — a tidal volume of 8 ml/kg
  Arms: Volume-controlled ventilation
Procedure: Pressure-controlled ventilation — a peak airway pressure to maintain a tidal volume of 8 ml/kg
  Arms: Pressure-controlled ventilation

SUMMARY:
Ischemia-reperfusion injury resulted from pneumoperitoneum during laparoscopic surgery have been reported in some literatures. There are no studies investigating the time course of changes in oxidative stress markers in volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) modes. The aim of this study is to compare the alterations in oxidative stress in two different ventilation strategies during gynecologic laparoscopic surgery.

Methods:

Fifty-two patients of ASA physical status I or II were randomly assigned to receive either VCV or PCV during laparoscopic gynecologic surgery. Blood gas analysis and ventilation variables were recorded 1 minute before (T1) and 1 hour after (T2) pneumoperitoneum. Blood samples for malondialdehyde (MDA) measurement were collected at seven points: 1 minute before (T1) and 1 hour after (T2) pneumoperitoneum; 30 minutes, 60 minutes, 90 minutes, and 120 minutes after deflation (T3~T6); and 24 hours after deflation (T7).

DETAILED DESCRIPTION:
Pneumoperitoneum during laparoscopic procedures greatly impairs splanchnic blood flow due to compression. Increased intra-abdominal pressure may elevate the diaphragm, increase intra-thoracic pressure, reduce functional residual capacity, and thus lead to atelectasis. In a collapsed lung, blood flow is decreased and reperfusion injury may subsequently occur during re-expansion of the lung. This ischemia-reperfusion injury results from the formation of reactive oxygen species (ROS), which are highly reactive intermediates of the oxygen metabolism. When there is an imbalance between ROS generation and removal by antioxidative mechanisms, oxidative stress occurs and eventually causes cellular and organ damage. Oxidative stress mediates tissue injury and may represent an important link between laparoscopy and clinical side effects. Malondialdehyde (MDA) is considered the most reliable marker of oxidative stress in the clinical setting. It is a breakdown product of lipid peroxidation in tissues. An elevated concentration of MDA reflects the level of lipid peroxidation.

Although there is abundant data comparing the effects of VCV and PCV during laparoscopic surgery, the time course of changes in oxidative stress in these two modes has not been elucidated. Therefore, the aim of this study was to compare the alterations of oxidative stress in two different ventilation modes, VCV and PCV, during gynecologic laparoscopic surgery. To this end, the investigators established a prospective randomized clinical study and measured the plasma levels of a lipid peroxidation marker at different stages.

Fifty-two patients of ASA physical status I or II were randomly assigned to receive either VCV or PCV during laparoscopic gynecologic surgery. During the operation, blood gas analysis and ventilation variables were recorded 1 minute before (T1) and 1 hour after (T2) the establishment of CO2 pneumoperitoneum in both groups. Blood samples for MDA measurement were collected at seven points: 1 minute before (T1) and 1 hour after (T2) pneumoperitoneum; at intervals of 30 minutes for 2 hours after the deflation of CO2 (T3~T6); and 24 hours after the deflation of CO2 (T7). The samples were immediately centrifuged (1000g, 10 minutes) and the supernatants were stored at -800C until further analysis, which took place within 1 week. The investigators assessed the quality of recovery from anesthesia using a nine-item quality of recovery score (QoR Score) before operation and 24 hours after the deflation of CO2.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 70 years with a BMI < 30 kg/m2 scheduled for laparoscopic gynecologic surgery requiring at least 1 hour of pneumoperitoneum

Exclusion Criteria:

* cardiopulmonary disease and a history of sepsis or shock, findings suspicious of malignant disease, previous major abdominal operation, smoking, and recent antioxidant use (i.e. vitamins A, C and E).

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
peak airway pressure | 1 hour after the establishment of CO2 pneumoperitoneum
  During surgery, CO2 pneumoperitoneum was induced with an intraabdominal pressure of 15 mmHg. After one hour of pneumoperitoneum, ventilation variables were recorded.

SECONDARY OUTCOMES:
plasma MDA concentration | 1 minute before (T1) and 1 hour after (T2) pneumoperitoneum; at intervals of 30 minutes for 2 hours after the deflation of CO2 (T3~T6); and 24 hours after the deflation of CO2 (T7)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chih Liao, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Anesthesiology, Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Background] Sammour T, Mittal A, Loveday BP, Kahokehr A, Phillips AR, Windsor JA, Hill AG. Systematic review of oxidative stress associated with pneumoperitoneum. Br J Surg. 2009 Aug;96(8):836-50. doi: 10.1002/bjs.6651. PMID 19591166
- [Background] Del Rio D, Stewart AJ, Pellegrini N. A review of recent studies on malondialdehyde as toxic molecule and biological marker of oxidative stress. Nutr Metab Cardiovasc Dis. 2005 Aug;15(4):316-28. doi: 10.1016/j.numecd.2005.05.003. PMID 16054557
- [Background] Kontoulis TM, Pissas DG, Pavlidis TE, Pissas GG, Lalountas MA, Koliakos G, Topouridou K, Sakantamis AK. The oxidative effect of prolonged CO(2) pneumoperitoneum a comparative study in rats. J Surg Res. 2012 Jun 15;175(2):259-64. doi: 10.1016/j.jss.2011.09.030. Epub 2011 Oct 12. PMID 22172128